CLINICAL TRIAL: NCT03059459
Title: Effect of Atmospheric Pollution Due to Particulate Matter on Obstructive Lung Diseases in San Nicolas, Buenos Aires Province, Argentina
Brief Title: Effect of Atmospheric Pollution on Obstructive Lung Diseases
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Council of Scientific and Technical Research, Argentina (Other Government)
Responsible Party: Principal Investigator, Pablo Orellano, Dr.PH, Researcher, National Council of Scientific and Technical Research, Argentina
Other Study IDs: 2919/1191/15
Record Dates: First submitted 2017-02-15; First posted 2017-02-23 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Lung Diseases, Obstructive
Keywords: Lung Diseases, Obstructive; Air Pollution; Particulate Matter
MeSH Terms: conditions — Lung Diseases, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Several studies have demonstrated the association between atmospheric pollution and chronic respiratory diseases. The magnitude of this association and its dependence of local factors are still unknown in Argentina, particularly for obstructive lung diseases like asthma and chronic obstructive pulmonary disease (COPD). The objective of this study is to assess the effect of atmospheric pollution due to particulate matter (PM) on asthma and COPD exacerbations in adults. A prospective cohort study will be carried out in patients attending the pulmonary service of a public hospital located in San Nicolas, Buenos Aires province, Argentina. Patients will be followed for 12 months after recruitment. The outcome variables will be the frequency of hospitalizations or emergency department consults for asthma or COPD exacerbations and related conditions, and the impact of COPD on a person's life as measured by the COPD assessment test (CAT) questionnaire. The exposure will be the pollution level in the particular address, measuring PM10 concentrations with portable equipment. Other variables as air temperature, humidity, and individual patient risk factors will be considered as potential confounders or effect modifiers. The associations will be estimated through regression models, i.e. logistic and Poisson regressions and recurrent event survival analysis. The results of this study should provide elements to estimate the risk of chronic respiratory diseases associated with atmospheric pollution, and to evaluate strategies for risk assessment in the local community.

ELIGIBILITY:
Inclusion Criteria:

* Patients with asthma or COPD attending the pulmonary service.

Exclusion Criteria:

* Patients who refuse to participate in this study or to sign the informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending the pulmonary service of a public hospital located in San Nicolas, Buenos Aires province, Argentina.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2015-12-04 (Actual); Primary Completion 2018-12-04 (Estimated); Study Completion 2018-12-04 (Estimated)

PRIMARY OUTCOMES:
Asthma or COPD hospitalizations or emergency department visits | 12 months
  Asthma or COPD hospitalizations or emergency department visits measured by hospital records

SECONDARY OUTCOMES:
Quality of life associated with obstructive lung diseases | 12 months
  The quality of life associated with obstructive lung diseases will be measured with a short patient-completed questionnaire, the COPD Assessment Test (CAT).

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Orellano, Dr.PH, Principal Investigator — National Scientific and Technical Research Council, Argentina

IPD SHARING:
Plan to Share IPD: No